CLINICAL TRIAL: NCT00541762
Title: Mechanistic Study (Physiology)
Brief Title: Regulation of Fat-stimulated Neurotensin Secretion in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EKBB 86/05; SNF Grant. 3200-065588.04/1
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Neurotensin; Human; Physiology of neurotensin; fat perfusion; healthy subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A, 3; B, 3; C, 3 (Other): A, 3: Fat with and without orlistat or placebo. B, 3: LCF vs MCF vs placebo. C, 3: LCF with and without DEXLOX or placebo.
  Interventions: Dietary Supplement: Fat perfusion to the small intestine

INTERVENTIONS:
Dietary Supplement: Fat perfusion to the small intestine — 1. Triglycerides, long chain fatty acids, medium chain fatty acids perfused to the small intestine
  2. Orlistat perfused to the small intestine
  3. DEXLOX as CCK-1 receptor antagonist

SUMMARY:
Context: Cholecystokinin (CCK) and neurotensin are stimulated during meal intake by the presence of fat in the small intestine. The sequence of events suggests that fat hydrolysis is crucial for triggering the release.

Objectives: The aim of this study was therefore to investigate whether CCK mediated the effect of intraduodenal (ID) fat on neurotensin secretion via CCK-1 receptors.

DETAILED DESCRIPTION:
Setting: Single center study; 34 male volunteers were studied in consecutive, randomized, double blind, crossover studies.

Subjects and Methods: CCK and neurotensin release were quantified in: 1) 12 subjects receiving an ID fat infusion with or without 60 mg orlistat, an irreversible inhibitor of gastrointestinal lipases, in comparison to vehicle. 2) 12 subjects receiving ID long chain fatty acids (LCF), ID medium chain fatty acids (MCF) or ID vehicle. 3) 10 subjects receiving ID LCF with and without the CCK-1 receptor antagonist dexloxiglumide (DEXLOX) or ID vehicle plus IV saline (placebo). Hormone concentrations were measured by specific RIA systems.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Neurotensin plasma concentrations | Change in plasma cocnentrations over 2-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Drewe, MD, Principal Investigator — University Hospital, 4031 Basel, Switzerland; Christoph Beglinger, MD, Principal Investigator — Department of Research and Clinical Pharmacology, University Hospital, Basel Switzerland
Locations (1):
- Clinical Research Center, University Hospital, Basel, Switzerland

REFERENCES:
- [Background] Ferris CF, Carraway RE, Hammer RA, Leeman SE. Release and degradation of neurotensin during perfusion of rat small intestine with lipid. Regul Pept. 1985 Oct;12(2):101-11. doi: 10.1016/0167-0115(85)90191-0. PMID 3840906
- See also: publication in JCEM — http://www.ncbi.nlm.nih.gov/pubmed/18303078